CLINICAL TRIAL: NCT04910399
Title: Evaluation of the Effect of Peptides and n-3 Polyunsaturated Fatty Acids (n-3 PUFAs) From a Blue Fish Hydrolysate on Memory in Healthy Elderly People : a Randomised, Placebo-controlled, Double-blind Study.
Brief Title: Development of an Innovative Health Ingredient From Marine By-products for the Healthy Aging
Acronym: BRAINBOOSTER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abyss Ingredients (Industry)
Collaborators: Laboratoire Nutrition et Neurobiologie intégrée (Unknown); University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: BRAINBOOSTER
Record Dates: First submitted 2021-05-14; First posted 2021-06-02 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Memory Impairment; Age-related Cognitive Decline
Keywords: Memory; Cognitive decline; Food supplement; Hydrolysate; Aging
MeSH Terms: conditions — Memory Disorders; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blue fish hydrolysate (Experimental): The test product is a food supplement named BrainBooster in our project. It is presented as a capsule containing a blue fish hydrolysate, containing peptides and n-3 polyunsaturated fatty acids.
  Interventions: Dietary Supplement: Blue fish hydrolysate
- Placebo (Placebo Comparator): The placebo is a capsule with same appearance and organoleptic properties as the active product, containing no active component.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Blue fish hydrolysate — The experimental product is a dietary supplement composed of a hydrolysate of fatty blue fish containing low molecular weight peptides and n-3 polyunsaturated fatty acids.
  One of the two study groups (28 volunteers) will take 4 capsules of the active product (blue fish hydrolysate), for 90 days.
  Each day the capsules will be taken as followed : 2 capsules in the morning and 2 capsules in the evening.
  Arms: Blue fish hydrolysate
Dietary Supplement: Placebo — The placebo product containing mainly maltodextrin is presented in the same form as the active product, so that people handling the product cannot distinguish between them. The placebo is flavoured in order to have a fishy smell just like the active product.
  One of the two study groups (28 volunteers) will take 4 capsules of placebo per day, for 90 days.Each day the capsules will be taken as followed : 2 capsules in the morning and 2 capsules in the evening.
  Arms: Placebo

SUMMARY:
This interventional, randomised, placebo-controlled and double-blind study aims to evaluate the effect of a dietary supplementation with a blue fish hydrolysate derived from marine by-products, containing peptides and n-3 polyunsaturated fatty acids, on cognitive performance in a healthy older population, between 60 and 73 years old, with lower memory performance.

DETAILED DESCRIPTION:
The main objective of this study is to evaluate the efficacy of a dietary supplementation with a hydrolysate derived from marine by-products compared to a placebo on the evolution of episodic memory at 3 months in healthy elderly people with lower memory performance.

The secondary objectives of this study are to evaluate the efficacy of a dietary supplementation with a hydrolysate derived from marine by-products compared to a placebo on the evolution at 3 months of verbal recognition memory, working memory, perceived stress level, biological markers of nutritional and hormonal status in healthy elderly people with lower memory performance. Finally, participants' satisfaction with the product will be assessed.

Participants have to take 4 capsules per day of the hydrolysate containing 770 mg (dose per capsule) or of the placebo for 90 days.

Participants will have a phone screening interview and will attend 5 visits to the Bordeaux University Hospital on the Neuro-Psychopharmacological Research Platform.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, aged between 60 and 73 years old (including age limits),
* BMI between 20 and 30 kg/m2,
* Not diagnosed with Alzheimer's disease and autonomous,
* 26 < MMSE <= 29,
* PAL TEA > 57,
* Affiliated with a social security plan,
* Able to understand the study and consent,
* Available to come to the 5 visits required for the study,
* Informed and have signed an informed consent.

Exclusion Criteria:

* Person who has participated in the last 3 months or is currently participating in another clinical trial that may interfere with the evaluation of the primary endpoint (memory).
* Subject consuming food supplements likely to have an effect on memory or within less than 6 months
* Subject consuming high level of Vitamin A and/or Long chain n-3 PUFA evaluated by a food frequency questionnaire
* Restrictive or unbalanced diet (hypocaloric, vegetarian, vegan, …) self-declared at V0
* Fish consumption more than twice a week
* Allergy to fish
* Life threatening pathology (such as cancer) in remission for less than 1 year or still ongoing,
* Diabetes (type 1 or type 2),
* Cardiovascular disease diagnosed within less that 2 years, with the following exceptions: subjects with controlled (medicated) high blood pressure and/ or controlled (medicated) can be included,
* Personal history of stroke
* Personal history of schizophrenia or other psychiatric disorders
* Ongoing neuroleptic treatment
* Current depressive episode characterized at clinical interview according to the criteria of module A of the MINI (Mini International Neuropsychiatric Interview)
* Unbalanced thyroid disease (treatment modified in the last 6 months),
* For women: hormone replacement therapy started less than 3 months ago or for which the dosage of the treatment has been modified in the last 3 months or whose dosage is likely to be modified during the study
* Chronic inflammatory bowel disease or chronic disorders of intestinal absorption
* Diagnosed inflammatory bowel disease or chronic intestinal absorption disorders
* Current antidepressant treatment or discontinuation within the last 3 months
* Substance abuse or alcoholism within the last 6 months (smoking is allowed)
* General anesthesia in the last 6 months or scheduled in the next 6 months
* Alcohol abuse: more than 2 standard drinks per day,
* Subjects with clinical characteristics that may interfere with the performance of the tests (e.g.: acute visual or hearing impairment)
* Person placed under court protection,
* Person participating in another research study with an exclusion period still in progress ongoing,

Ages: 60 Years to 73 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-08-10 (Actual)

PRIMARY OUTCOMES:
CANTAB - Paired Associate Learning test (PAL TEA = PAL Total Error Adjusted) | 12 weeks

SECONDARY OUTCOMES:
CANTAB - Paired Associate Learning test (PAL) | 12 weeks
CANTAB - Verbal Recognition Memory (VRM) | 12 weeks
CANTAB - Spatial Working Memory test (SWM) | 12 weeks
CANTAB - Spatial Span test (SSP) | 12 weeks
CANTAB - Reverse Spatial Span test (Reverse SSP) | 12 weeks
Perceived Stress Level Scale (PSS) | 12 weeks
  The Perceived Stress Scale is a 10-item self-administered questionnaire that assesses the frequency with which the respondent has experienced feelings of stress or loss of control over events in the past month. Each item is rated by the patient on a Likert scale from 0 to 4. The total score is obtained by adding the score for each item. The total score is between 0 and 40. A score below 13 suggests a low stress level, a score between 14 and 19 a moderate stress level and a score above 20 a high stress level.
Mini-Mental State Examination (MMSE) | 12 weeks
  The MMSE consists of 30 questions or tasks (items) exploring possible disorders of: orientation in time and space, memory, attention, language (speech, comprehension, reading, writing), motor performance. For each of the thirty questions, a correct answer results in a score of 1 and a wrong or approximate answer in a score of 0. The final score is marked out of 30 points.
Geriatric Depression Scale (GDS) | 12 weeks
  The GDS Short Form is a self-administered questionnaire with 15 items, each with a binary Yes-No response. It was designed to test for depressive symptoms in elderly subjects. In the original form of the scale, an individual with a score of 0 to 5 is considered normal. A score between 5 and 9 indicates a high probability of depression and a score between 10 and 15 almost always indicates depression.
Participant's Satisfaction via a multiple choice questionnaire | 12 weeks
  Each volunteer will filled a multiple choice questionnaire at the end of the study. The galenic choice, organoleptic aspects and the global intake of the product they took will be evaluated.

OTHER OUTCOMES:
Concentration of fasting blood glucose | baseline and 12 weeks
Concentration of fasting blood Total-cholesterol | baseline and 12 weeks
Concentration of fasting blood HDL-cholesterol | baseline and 12 weeks
Concentration of fasting blood LDL-cholesterol | baseline and 12 weeks
Concentration of fasting blood triglycerides | baseline and 12 weeks
Concentration of cytokines | baseline and 12 weeks
  An inflammatory marker in plasma
Concentration of oxylipins | baseline and 12 weeks
  An inflammatory marker in plasma
Concentration of salivary cortisol | baseline and 12 weeks
  Collection 30 minutes after awakening
Concentration of urinary cortisol | baseline and 12 weeks
  Collection after awakening
Concentration of urinary cortisol metabolites | baseline and 12 weeks
  Dosage of tetrahydrocortisone and tetrahydrocortisol. Collection after awakening

CONTACTS AND LOCATIONS:
Overall Officials: Pierre PHILIP, Pr, Principal Investigator — University Hospital, Bordeaux
Locations (2):
- France (2):
  - Laboratoire Nutrition et Neurobiologie Intégrée, Bordeaux
  - Plateforme de Recherche Neuro-Psychopharmacologique USR CNRS 3413 SANPSY, CHU de Bordeaux, Bordeaux